CLINICAL TRIAL: NCT04692909
Title: Deep Transcranial Magnetic Stimulation (dTMS) of the Medial Prefrontal Cortex (mPFC) in Food Addiction and Obesity
Brief Title: Deep Transcranial Magnetic Stimulation (dTMS) of the Medial Prefrontal Cortex in Food Addiction and Obesity
Acronym: FAOB-mPFC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOR032415CTIL
Record Dates: First submitted 2020-09-24; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-09

CONDITIONS: Food Addiction; Obesity, Morbid
MeSH Terms: conditions — Food Addiction; Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Active dTMS
  Interventions: Device: dTMS with mPFC stimulation
- Placebo (Placebo Comparator): Placebo dTMS
  Interventions: Device: dTMS with mPFC stimulation

INTERVENTIONS:
Device: dTMS with mPFC stimulation — dTMS with Brainsway's H7 device, stimulating the mPFC.

SUMMARY:
This experiment is based on a unique technique of deep Transcranial magnetic stimulation (dTMS) of the brain's cortex, aiming to produce weight loss in food-addicted severely obese adults.

DETAILED DESCRIPTION:
The neurobiological underpinnings of food addiction in obesity point to chemical, structural and functional imbalance in the mesolimbic dopaminergic brain system. This may cause symptoms of altered reward processing, excessive cravings for hyperpalatable food and repeated self-regulation failures to control food intake in this population. Specifically, the medial prefrontal cortex (mPFC), anterior cingulate cortex (ACC) and deeper reward-related brain regions function differentially from healthy controls and similarly to individuals with substance or behavioral addiction. Deep transcranial magnetic stimulation of the mPFC has been shown efficacious in reducing cravings and other addictive symptoms in individuals with SUD, as well as symptoms of compulsivity in obsessive compulsive disorder (OCD). In this study the investigators use deep transcranial magnetic stimulation (dTMS) with an H-coil to safely stimulate the mPFC and deeper brain regions, in individuals with obesity and food addiction. The investigators aim to produce neuroplasticity favoring the restoration of mPFC functioning, alleviating food addiction symptoms and promoting weight loss.

ELIGIBILITY:
Inclusion Criteria:

* 30 ≤ BMI ≥ 50.
* Having had at least one prior conventional weight loss attempt, but no current weight loss attempts or over the last 3 months.
* Having satisfied a safety screening questionnaire for TMS (Keel, 2001)
* Omnivorous
* Have not had experience with TMS of any kind
* Exclusion Criteria:
* They experience tremor in any limb.
* They experience seizures.
* They have a history of epilepsy or seizure (EXCEPT those therapeutically induced by ECT, or febrile childhood seizures).
* They are at increased risk for seizures for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or a history of significant head trauma with loss of consciousness for > 5 minutes.
* A history of clinically significant neurological disorders, including organic brain disease, epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery or personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes (self-reported history).
* They have a clinically significant hearing impairment, unless a medical letter is provided permitting the participant to receive a dTMS treatment.
* The participant has an unstable physical disease, such as acute unstable cardiac disease, or high blood pressure (>150 mmHg, systolic/> 110 mmHg diastolic, unless a medical letter is provided permitting the participant to receive a dTMS treatment.

Exclusion criteria:

* They experience tremor in any limb.
* They experience seizures.
* They have a history of epilepsy or seizure (EXCEPT those therapeutically induced by ECT, or febrile childhood seizures).
* They are at increased risk for seizures for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or a history of significant head trauma with loss of consciousness for > 5 minutes.
* A history of clinically significant neurological disorders, including organic brain disease, epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery or personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes (self-reported history).
* They have a clinically significant hearing impairment, unless a medical letter is provided permitting the participant to receive a dTMS treatment.
* The participant has an unstable physical disease, such as acute unstable cardiac disease, or high blood pressure (>150 mmHg, systolic/> 110 mmHg diastolic, unless a medical letter is provided permitting the participant to receive a dTMS treatment.
* The participant is at a high risk for severe violence or suicidal tendencies, has current DSM5 diagnosis of schizophrenia, bipolar disorder, or other psychotic disorder, as reported during the screening interview (see appendix 3).
* The participant has metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neuro-stimulators, intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or implanted medical pumps.
* The participant is having, or has had, any metal in the head (outside the mouth).
* The participant has any cognitive or functional disability, according to criteria specified in the DSM-V, such as active and unstable psychiatric disorder according to DSM-V (Axis I and Axis II), diagnosed within the last year.
* The participant has started or changed a psychotropic prescription within the past three months.
* The participant has current alcohol or other substance abuse or dependence, or has had one over the past 12 months prior to recruitment.
* The participant can't reliably communicate with the investigator, or is unlikely to cope with the requirements of the experiment.
* The participant is having a known or suspected pregnancy or lactation.
* The motor threshold can't be found or quantified.
* The PI decides that the participant should be withdrawn from the study for the safety and welfare of the participant. For example, the participant experiences adverse event which is contraindicated with the continuation in the study.
* The participant has a history of intolerance to a TMS treatment. The participant asks for withdrawal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in BMI | Change in BMI between baseline and the end of the treatment (day 15) and follow-up (a month after day 15)
  Unit of measure: BMI in kg/m^2 (weight in kilograms, height in meters)
Change in BMI | Change in BMI between baseline and follow-up (a month after day 15)
  Unit of measure: BMI in kg/m^2 (weight in kilograms, height in meters)

SECONDARY OUTCOMES:
Change in food addiction symptoms on the Yale Food Addiction Scale (YFAS) | The change in the number of symptoms on day 15 compared to baseline will be assessed.
  The YFAS includes 1-7 symptoms, while participants are recruited to the study if they have 3 symptoms or more. The greater the symptoms, the more food addiction the participants experience.
Change in food addiction symptoms on the Yale Food Addiction Scale (YFAS) | The change in the number of symptoms on day 16 (a month after day 15) compared to baseline will be assessed.
  The YFAS includes 1-7 symptoms, while participants are recruited to the study if they have 3 symptoms or more. The greater the symptoms, the more food addiction the participants experience.
Cognitive regulation of eating | The change in reaction time on the Food Stroop task between day 15 and baseline.
  Cognitive regulation of eating will be assessed with a computerized Food Stroop task. A change in reaction time (milliseconds) in response to high-calorie food, low-calorie food, and non-food items will be assessed.
Cognitive regulation of eating | The change in reaction time on the Food Stroop task between day 16 (a month after day 15) and baseline.
  Cognitive regulation of eating will be assessed with a computerized Food Stroop task. A change in reaction time (milliseconds) in response to high-calorie food, low-calorie food, and non-food items will be assessed.
Depressive symptoms | A change in BDI score from baseline to day 15.
  Depressive symptoms will be assessed with the 21-question multiple-choice self-report inventory, the Beck Depression Inventory (BDI). The highest possible total for the whole test would be sixty-three and the lowest possible score for the test would be zero.
Depressive symptoms | A change in BDI score from baseline to day 16.
  Depressive symptoms will be assessed with the 21-question multiple-choice self-report inventory, the Beck Depression Inventory (BDI). The highest possible total for the whole test would be sixty-three and the lowest possible score for the test would be zero.
Eating behavior [cognitive restraint (CR), emotional eating (EE), uncontrollable eating (UE)] will be assessed with the Three Factor Eating Questionnaire (TFEQ). | The change in these parameters will be assessed between baseline and day 15.
  The TFEQ measures CR, EE, and UE. A change (decrease or increase) in the symptoms of each of the scales will be assessed at the end of the intervention and at follow up.
Eating behavior [cognitive restraint (CR), emotional eating (EE), uncontrollable eating (UE)] will be assessed with the Three Factor Eating Questionnaire (TFEQ). | The change in these parameters will be assessed between day 16 (a month after day 15) and baseline.
  The TFEQ measures CR, EE, and UE. A change (decrease or increase) in the symptoms of each of the scales will be assessed at the end of the intervention and at follow up.
Eating behavior [restrictive eating (RE), emotional eating (EME), external eating (EXE)] will be assessed with the Dutch Eating Behavior Questionnaire (DEBQ) | The change in these parameters will be assessed between baseline and day 15.
  The DEBQ measures RE, EME and EXE, A change (decrease or increase) in the symptoms of each of the scales will be assessed at the end of the intervention and at follow up.
Eating behavior [restrictive eating (RE), emotional eating (EME), external eating (EXE)] | The change in these parameters will be assessed between day 16 (a month after day 15) and baseline.
  The DEBQ measures RE, EME and EXE, A change (decrease or increase) in the
Binge eating frequency | The change in binge eating frequency between baseline and day 15.
  Binge eating will be assessed with the Eating disorder examination-questionnaire with Instructions (EDE-Q-I). This questionnaire assesses binge eating frequency over the past 28 days.
Binge eating frequency | The change in binge eating frequency between baseline and day 16.
  Binge eating will be assessed with the Eating disorder examination-questionnaire with Instructions (EDE-Q-I). This questionnaire assesses binge eating frequency over the past 28 days.
Quality of life | The change in the SF-36 score between baseline and day 15.
  Health Status Scale Short-form 36 (SF-36)
Quality of life | The change in the SF-36 score between baseline and day 16.
  Health Status Scale Short-form 36 (SF-36)
General mood | The change in the overall score (positive affect minus negative affect) between baseline and day 15.
  Positive Affect Negative Affect Schedule (PANAS).
General mood | The change in the overall score (positive affect minus negative affect) between baseline and day 16.
  Positive Affect Negative Affect Schedule (PANAS).

CONTACTS AND LOCATIONS:
Overall Officials: Roni Aviram-Friedman, PhD, Study Director — Ben-Gurion University of the Negev
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: Undecided